CLINICAL TRIAL: NCT01418274
Title: A Study to Investigate the Effect of Multiple Doses of Danoprevir/Ritonavir (DNV/RTV) on the Pharmacokinetics (PK) of Escitalopram (ESC) and S-Demethylcitalopram (S-DCT) in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Danoprevir/Ritonavir on the Pharmacokinetics of Escitalopram and S-Demethylcitalopram in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP25643
Record Dates: First submitted 2011-07-20; First posted 2011-08-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — danoprevir; Escitalopram; Ritonavir

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: danoprevir; Drug: escitalopram; Drug: ritonavir

INTERVENTIONS:
Drug: danoprevir — oral doses of danoprevir
Drug: escitalopram — oral doses of escitalopram
Drug: ritonavir — oral doses of ritonavir

SUMMARY:
This single-arm, open-label, non-randomized study will evaluate the effect of danoprevir/ritonavir on the pharmacokinetics of escitalopram and S-demethylcitalopram in healthy volunteers. Healthy volunteers will receive oral doses of danoprevir/ritonavir and escitalopram. The anticipated time of the study is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers, aged 18 to 55 years, inclusive
* Body mass index (BMI) 18.0 to 32.0 kg, inclusive
* Absence of evidence of any active or chronic disease
* Non-smokers

Exclusion Criteria:

* Presence of any active or chronic disease
* Abnormal blood pressure
* Abnormal resting heart rate
* Abnormal ECG values
* History of any clinically significant cardiovascular or cerebrovascular disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in area under the plasma concentration time curve (AUC) of escitalopram | Approximately 4 weeks

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | Approximately 6 weeks
Effect on pharmacokinetics of major escitalopram metabolite: change in AUC of S-demethylcitalopram | Approximately 4 weeks
Effect of co-administration of escitalopram on danoprevir/ritonavir steady-state pharmacokinetics: change in AUC of danoprevir/ritonavir | Approximately 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Lenexa, Kansas, United States